CLINICAL TRIAL: NCT03206112
Title: Loss of Depotentiation in Focal Dystonia
Status: Terminated | Type: Observational
Why Stopped: PI leaving the NIH
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170123; 17-N-0123
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Focal Dystonia; Healthy Volunteers
Keywords: Focal Dystonia; Healthy Volunteers; Paired Associative Stimulation (PAS)
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focal Dystonia: Subjects diagnosed with Focal Dystonia
  Interventions: Other: PAS25; Other: PAS10; Other: PAS25-cTBS150
- Healthy Volunteers: Healthy Volunteers
  Interventions: Other: PAS25; Other: PAS10; Other: PAS25-cTBS150

INTERVENTIONS:
Other: PAS25 — We will record surface electromyography from the target abductor pollicis brevis muscle and adjacent first dorsal interosseous and abductor digiti minimi muscles.
Other: PAS10 — We will record surface electromyography from the target abductor pollicis brevis muscle and adjacent first dorsal interosseous and abductor digiti minimi muscles. TBS is a special form of
Other: PAS25-cTBS150 — We will record surface electromyography from the target abductor pollicis brevis muscle and adjacent first dorsal interosseous and abductor digiti minimi muscles.

SUMMARY:
Background

Focal dystonia is a brain disorder. It affects a muscle or muscles in a specific part of the body. Researchers think it may be related to excessive training or practice. They want to know more about how much training might trigger focal dystonia.

Objectives:

To study why people develop focal dystonia. To study how brain plasticity changes with focal dystonia.

Eligibility:

People at least 18 years of age with focal dystonia.

Healthy volunteers the same age are also needed.

Design:

Participants will be screened with a physical exam and questions. They may have blood and urine tests.

Participants will have up to 3 testing visits.

Participants will have small electrodes stuck on the skin on the hands or arms. Muscle activity will be recorded.

Participants will have transcranial magnetic stimulation (TMS). A wire coil will be placed onto the scalp. A brief electrical current will pass through the coil. The current will create a magnetic field that affects brain activity.

Participants may be asked to tense certain muscles or do simple actions during TMS.

A nerve at the wrist will get weak electrical stimulation. The stimulation may be paired with TMS for very short times.

Participants will receive repeated magnetic pulses. Participants will receive a total of 150 pulses during a 10-second period. An entire testing visit will last about 3 hours.

...

DETAILED DESCRIPTION:
Objectives

Simulation paradigms can induce plastic changes in brain excitability. Paired associative stimulation (PAS) with an interstimulus interval of 25 ms (PAS25) induces a long-term potentiation (LTP)-like effect while that at an interval of 10 ms (PAS10) induces a long-term depression (LTD)-like effect. The LTP-like effect induced by PAS25 is exaggerated in patients with focal dystonia. The LTD-like effect with PAS10 is also increased in focal dystonia but not in the target area of PAS. Depotentiation refers to the reversal of LTP by which LTP is abolished by a following procedure that has no effect when it is given alone. Brain-derived neurotrophic factor has a variety of roles in modulating both LTP and LTD. The Val66Met single nucleotide polymorphism is related to abnormal cortical plasticity. In this protocol, we propose a study to test the hypothesis that depotentiation is weaker in focal dystonia patients compared to healthy controls. In addition, motor cortical inhibition is decreased in focal dystonia. We will test the changes in motor cortical inhibition following different interventional procedures in focal dystonia. We will also test the relationship between depotentiation and LTP/LTD-like effects in focal dystonia patients.

Study population

We intend to study up to 20 patients with focal dystonia and 20 age-matched healthy volunteers. Subjects will complete up to 3 study visits involving 3 different interventional procedures. Various outcome measures will be performed during each study visit.

Design

This is a hypothesis-driven study. We will compare the depotentiation effect in patients with focal dystonia to that in healthy volunteers. Patients will be evaluated with a clinical rating scale during the screening visit. Three interventional procedures will be tested during three study visits. Specifically, PAS25-cTBS150 tests the primary hypothesis with a depotentiation effect. PAS25 tests LTP-like effect and PAS10 tests the LTD-like effect. We will investigate the difference in outcome measures between patients and healthy volunteers after the interventional procedures. We will perform genetic tests to identify the brain-derived neurotrophic factor genotype in the patients and healthy volunteers.

Outcome measures

The primary outcome measure is motor-evoked potential (MEP) induced by transcranial magnetic stimulation immediately after the interventional procedure of PAS25-cTBS150. We will compare MEP amplitude in patients with that in healthy volunteers to identify whether depotentiation is weaker in focal dystonia. The secondary outcome measures are MEP amplitudes at other time points after the PAS25-cTBS150 procedure. We will also perform exploratory studies to investigate the effects of interventional procedures of PAS25 and PAS10 alone. We will test the relationship between depotentiation and LTP/LTD-like effects in focal dystonia. We will also study other exploratory outcome measures such as: resting and active motor threshold, MEP recruitment curve, excitability of motor cortical circuits (short- and long-interval intracortical inhibition, and intracortical facilitation) after three different interventional procedures.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for healthy controls:

* At least 18 years old.*
* Able to give informed consent.
* Able to comply with all study procedures.
* Abstain from alcohol for at least 48 hours prior to each study visit and caffeine on the day of the visit.
* Have no neurological or psychiatric disorders established by history and physical/neurological examination.

  * = A maximum of 10 subjects who are over the age of 70 will be screened for plasticity. If none of these subjects have plasticity, we will not accrue any more subjects over the age of 70.

Inclusion criteria for focal dystonia patients:

* At least 18-years old.*
* Able to give informed consent.
* Able to comply with all study procedures.
* Abstain from alcohol for at least 48 hours prior to each visit of the study and caffeine on the day of the visit.
* Have an established diagnosis of focal dystonia.
* No botulinum toxin injections at least in the past 3 months.

  * = A maximum of 10 subjects who are over the age of 70 will be screened for plasticity. If none of these subjects have plasticity, we will not accrue any more subjects over the age of 70.

EXCLUSION CRITERIA:

* Self-reported consumption of > 14 alcoholic drinks/week for a man and > 7 alcoholic drinks/week for a woman.
* Focal dystonia patients: presence of abnormal findings on neurological examination except for the diagnosis of focal dystonia. Healthy volunteers: no abnormal findings on neurological examination.
* History of or current brain tumor, stroke, head trauma with loss of consciousness, epilepsy or seizures.
* Have a Baclofen pump, or have neurostimulators for pain.
* Pregnant or breastfeeding women.
* Current episode of major depression or any major psychiatric illness.
* Presence of any metal in the eye or skull area such as a brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, metal fragments in the eye.
* Presence of pacemaker, intracardiac lines, implanted pumps or stimulators.
* Known hearing loss.
* Cognitive impairment.
* NIH staff from HMCS.

Healthy Volunteers:

-Taking medications that act directly on the central nervous system such as anti- epileptics, anti-histamines, anti-parkinsonian medication, medication for insomnia, anti-depressants, anti-anxiety medication.

Focal Dystonia Patients:

-Taking medications that act directly on the central nervous system such as anti- epileptics, anti-parkinsonian medication, medication for insomnia.

NOTE: Patients taking anti-histamines, anti-depressants or anti-anxiety medications will not be excluded from the protocol. However, only patients who have mild symptoms and agree to temporarily stop the medications during the experiment will be included.

Patients with mild symptoms of depression will be confirmed using Hamilton Depression Rating Scale with total scores below 13. Patients with mild symptoms of anxiety will be confirmed using Hamilton Anxiety Rating Scale with total scores below 17. Patients will be required to stop their medication at least 5 half- lives of the drug, but no longer than 5 days (even if the half-life is longer than 24 hours) before each experimental session.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects (patients and healthy volunteers) are recruited through the NIH Patient Recruitment and Public Liaison Office and from individuals who have participated in prior studies and are interested in being contacted for additional studies. Additionally, individuals who have contacted NIH to volunteer for research studies will be considered for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
MEP amplitude immediately after the PAS25-cTBS150 (depotentiation) protocol | throughout
  compare MEP amplitude in patients with that in healthy volunteers to identify whether depotentiation is weaker in focal dystonia

SECONDARY OUTCOMES:
MEP amplitudes | throughout
  MEP amplitudes at other time points after the PAS25-cTBS150 procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-N-0123.html